CLINICAL TRIAL: NCT06182774
Title: A Phase III Non-Inferiority Randomized Controlled Trial of Fixed Duration Versus Continuous Daratumumab Among Transplant Ineligible Older Adults With Newly Diagnosed Multiple Myeloma
Brief Title: Fixed Duration vs Continuous Daratumumab in Transplant Ineligible Older Adults With Newly Diagnosed Multiple Myeloma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Myeloma Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY13
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide; Dexamethasone; isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenalidomide & Dexamethasone (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- Daratumumab, Lenalidomide, Dexamethasone & Isatuximab (Active Comparator): Standard of Care
  Interventions: Drug: Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Isatuximab

INTERVENTIONS:
Drug: Daratumumab — Dose determined at enrollment
  Arms: Daratumumab, Lenalidomide, Dexamethasone & Isatuximab
Drug: Lenalidomide — Dose determined at enrollment
Drug: Dexamethasone — Dose determined at enrollment
Drug: Isatuximab — Dose determined at enrollment
  Arms: Daratumumab, Lenalidomide, Dexamethasone & Isatuximab

SUMMARY:
Currently, daratumumab or isatuximab are given continuously (non-stop), along side lenalidomide, and dexamethasone as part of multiple myeloma treatment. are given continuously (non-stop). Recent observations suggest that stopping daratumumab or isatuximb after about a year and a half of treatment may work just as well as giving them continuously with lenalidomide and dexamethasone. Sometimes, bortezomib is also given. This study is being done to answer the question: is less daratumumab or isatuximab treatment as good as more?

DETAILED DESCRIPTION:
The usual approach for people with myeloma who are not having a stem cell transplant is treatment with daratumumab or isatuximab in combination with lenalidomide, and dexamethasone. These drugs are given continuously until they are no longer effective or cause major side effects.

Those that decide to take part in this study, will be randomly placed in one of two groups. If in the usual care group, patients will continue all the myeloma medicines currently being taken. If in the experimental group, patients will stop the daratumumab or isatuximab injection, and continue taking the myeloma tablets currently being taken. Regardless of which group, patients will stay on treatment indefinitely as long they are benefiting from it.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed multiple myeloma that are transplant-ineligible
* Measurable disease at the time of diagnosis, as defined by at least one of the following criteria: Serum monoclonal protein (M-protein) ≥ 5 g/L; Urine M-protein ≥ 200 mg/24 hours; Involved serum free light chain measurement ≥ 100 mg/L, provided serum FLC ration is abnormal; For IgA patients whose disease can only be reliably measured by serum quantitative immunoglobulin ≥ 750 mg/dL
* Completed 18-20 cycles of daratumumab-lenalidomide-dexamethasone or isatuximab-lenalidomide-dexamethasone.
* Obtained at least a partial response per the standard 2016 IMWG criteria
* ECOG performance status 0-3
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life and/or health utility questionnaires in English, French, or a provided validated language.
* Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Participants must be accessible for treatment and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of participant enrollment.
* Participants of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Known history of concurrent amyloid light chain amyloidosis, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), and Waldenstrom's macroglobulinemia.
* Patients receiving concurrent treatment with other anti-cancer therapy that would impact the ability to comply with protocol treatment are ineligible. Note: Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of protocol treatment are eligible for this trial
* Active, uncontrolled bacterial, fungal, or viral infection within 7 days prior to enrollment.
* Known human immunodeficiency virus (HIV) with CD4 count < 350 cells/microliter. Note that patients who are HIV positive are eligible, provided:

  * They are under treatment with antiretroviral therapy for at least 4 weeks prior to enrollment, with acceptable pharmacokinetic interactions and minimal overlapping toxicity with protocol therapy AND
  * HIV viral load must be < 400 copies/ml within 16 weeks prior to enrollment AND
  * No history of opportunistic infections within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2032-01-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 9.1 years
  PFS is defined as the time from date of enrollment to date of first documentation of disease progression

SECONDARY OUTCOMES:
Overall Survival | 9.1 years
  Time from enrollment to death from any cause
Partial Response or Better as assessed by IMWG Criteria | 9.1 years
Incidence of Treatment-Related Grade 3-5 Adverse Events and all infections based on CTCAE 5.0 | 9.1 years
Time to Next Treatment | 9.1 years
  Time from enrollment to the start of next-line treatment
Post-protocol Therapy Documentation checklist | 9.1 years
  Documentation of patients 2nd line treatment after treatment completion of daratumumab, or isatuximab, lenalidomide, and dexamethasone
Quality of Life Utilizing EORTC QLQ-C30 | 9.1 years
Quality of Life Utilizing FACIT-COST | 9.1 years
Health Economic Analyses Utilizing EQ-5D-5L | 9.1 years
  Value is calculated by determining the incremental costs and benefits (life years, quality adjusted life years) across the two treatment arms from two perspectives, a health system and a societal perspective

CONTACTS AND LOCATIONS:
Overall Officials: Hira Mian, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario Canada
Locations (26):
- Canada (26):
  - BCCA - Kelowna, Kelowna, British Columbia
  - BCCA - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System, Brampton, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network (WRHN), Kitchener, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CIUSSS de l'Est-de-I'lle-de-Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data may be shared once the final analysis is complete following the Canadian Cancer Trials Group Data Sharing Policy available at https://ctg.queensu.ca/
URL: http://ctg.queensu.ca/